CLINICAL TRIAL: NCT05975970
Title: A Patient-Driven Augmented Reality-Based Rehabilitation System to Improve Upper Limb Amputee Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infinite Biomedical Technologies (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Alberta (Other)
Responsible Party: Principal Investigator, Rahul Kaliki, Chief Executive Officer, Infinite Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: W81XWH2010919
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Amputation; Upper Limb
Keywords: amputation; upper limb; myoelectric; training; prosthesis; augmented reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyoTrain AR System (Experimental): Participants will undergo functional task training using the MyoTrain AR system, which includes the HoloLens 2 augmented reality head-mounted display, four HTC VIVE SteamVR kinematic trackers, eight surface EMG electrodes based on the Element hardware platform, and a desktop computer. Participants will be prompted to use a pattern recognition-based myoelectric controller to operate a virtual prosthesis and complete a simulation of the GaMA Cup Transfer Task.
  Interventions: Device: MyoTrain AR
- Conventional Motor Imagery (Active Comparator): Participants will be provided motor imagery exercises that involve brief attempts to move the missing limb in a similar manner to how they would control their pattern recognition system to strengthen their muscles. These exercises do not involve any real-time control feedback or functional assessment.
  Interventions: Behavioral: Motor Imagery

INTERVENTIONS:
Device: MyoTrain AR — MyoTrain AR is a virtual prosthesis functional training system. From a hardware perspective it consists of an augmented reality head-mounted display (HMD), four SteamVR kinematic trackers, eight surface EMG electrodes based on the Element electrode platform, and a desktop computer to facilitate wireless communication between the various hardware components. From a software perspective, MyoTrain AR was developed in the cross-platform Unity 4.0 game development engine.
  Arms: MyoTrain AR System
Behavioral: Motor Imagery — Motor imagery describes the process by which a prosthesis user mentally simulates the execution of a desired limb movement and activates the musculature of the residual limb that would generate the desired movement.
  Arms: Conventional Motor Imagery

SUMMARY:
The investigators propose to evaluate the efficacy of MyoTrain AR in a prospective clinical study involving 10 individuals with trans-radial upper-limb loss over a period of 35 days. These individuals will be randomized to Group A (Control Group using conventional motor imagery exercises) and Group B (who will train with the MyoTrain AR system pre-prosthetically).

The investigators will test the following hypothesis: Pre-prosthetic training with the MyoTrain AR system, as compared to the current standard of care with conventional motor imagery exercises, results in improved subsequent control stability with the prosthesis.

Following a baseline functional assessment, participants will undergo a 30-day pre-prosthetic training period specific to their assigned Group. After this training period, participants will repeat the functional assessment. Participants will then receive their prosthetic device and occupational therapy consistent with the current clinical care standard, after which they will again undergo a battery of validated, clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Trans-radial unilateral limb loss with a healed residual limb
* Candidate for a 2+ degree-of-freedom (DoF) myoelectric pattern recognition prosthesis as determined by the study prosthetist
* Fluent in English
* Age of 18 years or greater

Exclusion Criteria:

* Prior experience with pattern recognition control
* Patients with a residual limb that is unhealed from the amputation surgery
* Patients with easily damaged or sensitive skin who would not tolerate EMG electrodes
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impactive full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
GaMA Cup Transfer Task Mean Completion Time | Day 35
  The time to successfully complete the entire task trial (all 4 cup movements) from start to finish; averaged over all successful trials.
GaMA Cup Transfer Task Mean Relative Grasp Duration | Day 35
  The percentage time spent in grasp phase relative to the entire movement (each movement involves reach-grasp-transport-release phases). This measure compensates for the expected inter-relation of absolute grasp duration with overall time, specifically identifying if grasp (object handling) is the main culprit in overall prolonged movement times.

SECONDARY OUTCOMES:
Assessment of Capacity for Myoelectric Controls (ACMC) | Day 35
  In contrast to other instruments, the ACMC does not require a specific set of tools or tasks. Instead, the proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. This outcome measure permits evaluation of bimanual tasks as well as different planes and work spaces of prosthesis use.
GaMA Cup Transfer Task Completion Rate | Day 35
  Percentage of successful trials out of 10 attempts. Note that errors (unsuccessful trials) may include not grasping the cup, or dropping or crushing the cup while in transport. This metric is therefore a general (non-specific) indication of grasp stability throughout the functional task. Errors other than grasp stability can result in an unsuccessful trial (hitting the barrier during transport, knocking a cup over during release, performing task in the wrong sequence) therefore type of error will also be tracked.
GaMA Cup Transfer Task Wrist Activation | Day 35
  The ability to coordinate two DoF (hand + wrist movements) is measured by the degree of active wrist rotation from neutral (starting) position at the time of grasp initiation. This measure will identify if there is coordinated use of wrist rotation at the appropriate movement time (at the end of the reach phase) in order to facilitate grasp.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No